CLINICAL TRIAL: NCT01010425
Title: Dose-ascending, Safety and Tolerability, Pharmacokinetic, and Pharmacodynamic Study of ACP-001 (TransCon PEG hGH)
Brief Title: Pharmacokinetics and Pharmacodynamics of ACP-001 (TransCon PEG hGH)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Study Director, Ascendis Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACP-001 (Prot. 3695)
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
MeSH Terms: interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACP-001, dose-level 1 (Experimental)
  Interventions: Drug: ACP-001 (TransCon PEG hGH); Drug: Placebo; Drug: Human Growth Hormone
- ACP-001, dose-level 2 (Experimental)
  Interventions: Drug: ACP-001 (TransCon PEG hGH); Drug: Placebo; Drug: Human Growth Hormone
- ACP-001, dose-level 3 (Experimental)
  Interventions: Drug: ACP-001 (TransCon PEG hGH); Drug: Placebo; Drug: Human Growth Hormone
- ACP-001, dose-level 4 (Experimental)
  Interventions: Drug: ACP-001 (TransCon PEG hGH); Drug: Placebo; Drug: Human Growth Hormone

INTERVENTIONS:
Drug: ACP-001 (TransCon PEG hGH) — ACP-001, dose-level 1, s.c., single-dose
  Arms: ACP-001, dose-level 1
Drug: ACP-001 (TransCon PEG hGH) — ACP-001, dose-level 2, s.c., single-dose
  Arms: ACP-001, dose-level 2
Drug: ACP-001 (TransCon PEG hGH) — ACP-001, dose-level 3, s.c., single-dose
  Arms: ACP-001, dose-level 3
Drug: ACP-001 (TransCon PEG hGH) — ACP-001, dose-level 4, s.c., single-dose
  Arms: ACP-001, dose-level 4
Drug: Placebo — Placebo, s.c., single-dose
Drug: Human Growth Hormone — Human Growth Hormone, s.c., daily for 7 days

SUMMARY:
Double-blind, randomized, placebo and active controlled dose-ascending study to investigate safety, tolerability, pharmacokinetics and pharmacodynamics of ACP-001 (TransCon PEG hGH).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* 20 to 45 years old
* Body Mass Index of 18.5 kg/m2 and less than or equal to 29.9 kg/m2
* Others

Exclusion Criteria:

* Known history of hypersensitivity to human growth hormone (hGH)
* Known history of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, immunological, hepatic or renal disease, or malignancies
* Others

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (adverse events, local reactions, immunogenicity) | 0-42 days
Pharmacokinetics; AUC and Cmax for hGH, TransCon-PEG hGH; and Pharmacodynamics measured by IGF-1 and IFG-BP | 0-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Ascendis Pharma, Study Director — Ascendis Pharma A/S
Locations (1):
- Toronto, Ontario, Canada

REFERENCES:
- [Derived] Gilfoyle D, Mortensen E, Christoffersen ED, Leff JA, Beckert M. A first-in-man phase 1 trial for long-acting TransCon Growth Hormone. Growth Horm IGF Res. 2018 Apr;39:34-39. doi: 10.1016/j.ghir.2017.12.002. Epub 2017 Dec 5. PMID 29273485